CLINICAL TRIAL: NCT03889301
Title: ¡Yo no Estoy Loc@! Improving Treatment Engagement for Latinos Using an E-E Video
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Collaborators: University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1228113-1
Record Dates: First submitted 2019-03-20; First posted 2019-03-26 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Anxiety Depression

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to experimental or control group.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-E Video (Experimental): Watch E-E video that incorporates health and educational messages
  Interventions: Behavioral: E-E Video
- Discussion (Active Comparator): Structured discussion about depression and anxiety
  Interventions: Behavioral: Discussion

INTERVENTIONS:
Behavioral: E-E Video — The E-E video was developed by the research team and chronicles the story of Ana who while enjoying coffee with two family members, shares her challenges with depression and her successful outcome with therapy. The video utilizes the genre of the telenovela which creates an entertaining environment where the audience is captivated by the content and absorbs the messages portrayed.
  Arms: E-E Video
Behavioral: Discussion — Structured psychoeducation and pamphlet about anxiety and depression.
  Arms: Discussion

SUMMARY:
The underutilization of behavioral health services for mood and anxiety disorders by Latinos is a public health concern warranting intervention development. Perceived stigma associated with the pursuit of behavioral health services disproportionately restricts mental healthcare in Latinos. The current study empirically tests an intervention aimed at improving perceptions of behavioral health services for mood and anxiety disorders, ultimately improving Latinos' mental health through access to treatment. The experimental intervention is based on the Entertainment-Education (E-E) model, a popular media campaign that incorporates health and educational messages in an entertaining, story-telling narrative. The E-E model incorporates characters who have characteristics, beliefs, attitudes, and behaviors that are similar to those of the targeted audience to maximize social validity. Using data gathered in focus groups with Latinos a 3-minute E-E video (in Spanish) that aims to reduce stigma towards mental illness and behavioral health services was developed. Sixty adult Latinos pursuing care at a Federally Qualified Health Center, who screen positive for anxiety and/or depression will be invited to participate in the study. Participants will be administered a structured demographic interview and measures that assess stigma and attitudes towards mental health and behavioral health services and then randomized to the E-E video or control (structured discussion about depression and anxiety) condition. Participants will then complete the study measures and be invited to attend a Cognitive Behavior Therapy (CBT) group for depression or anxiety. Consumer satisfaction will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Spanish-speaking

Exclusion Criteria:

* Screen positive for suicidality or psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Change in score on Generalized Anxiety Stigma Scale (GASS) | immediately before and immediately after intervention
  The GASS is a twenty-item scale used to measure stigma associated with anxiety disorders and was developed by Griffiths et al, (2004). It consists of two subscales, which measure two different types of stigma: personal and perceived. Responses to each item are measured on a five-point scale ranging from strongly disagree (0) to strongly agree (4). Scores on each subscale can range from 0 to 40. Higher scores indicate higher levels of stigma against generalized anxiety. A Spanish-language version of the measure is being tested for validity and reliability (Benuto & Gonzalez, In Progress).
Change in score on Depression Stigma Scale (DSS) | immediately before and immediately after intervention
  The DSS is an eighteen-item scale used to measure stigma associated with depression and was developed by Griffiths et al, (2004). It consists of two subscales, which measure two different types of stigma: personal and perceived. Responses to each item are measured on a five-point scale ranging from strongly disagree (0) to strongly agree (4).Scores on each subscale can range from 0 to 36. Higher scores indicate higher levels of stigma against depression. A Spanish-language version of the measure is being tested for validity and reliability (Benuto & Gonzalez, In Progress).
Change in score on Attitudes Towards Seeking Professional Help Scale (ATSPH) | immediately before and immediately after intervention
  The ATSPH is a 20-item item measure that is intended to reflect an individual's attitude toward professional behavioral health treatment. It is a modified version of the Attitudes Towards Seeking Professional Psychological Help Scale (Fisher & Turner, 1970). Responses to each item are measured on a four-point scale ranging from disagree (0) to agree (3). Items (including some that are reverse-scored) are summed; total scores can range from 0 to 30. Higher scores indicate more positive attitudes toward seeking treatment. A Spanish-language version of the measure is being tested for validity and reliability among a sample of Spanish-speaking individuals (Benuto & Gonzalez, In Progress).

CONTACTS AND LOCATIONS:
Locations (1):
- Community Health Alliance, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No